CLINICAL TRIAL: NCT05578417
Title: Treatment and Outcomes of Patients Identified With Non-Histaminergic Angioedema With Normal C1 Inhibitor in Canada
Brief Title: A Study to Review the Treatment and Outcomes of Teenagers and Adults With Non-histaminergic Angioedema With Normal C1 Inhibitor in Canada
Acronym: PROSPECT
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4013
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Hereditary Angioedema (HAE); Angioedema
Keywords: Drug Therapy
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HAE nC1-INH: Participants with HAE nC1-INH will be observed retrospectively for the treatments they receive and their outcomes in the real-world setting from January 1, 2012, to January 1, 2022.
  Interventions: Other: No Intervention
- NHAE nC1-INH: Participants with NHAE nC1-INH will be observed retrospectively for the treatments they receive and their outcomes in the real-world setting from January 1, 2012, to January 1, 2022.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
The main aim of this study is to describe the characteristics of participants, check for number of hereditary angioedema (HAE) cases, their treatment and outcomes. Another aim is to check how the healthcare facilities were utilized for treatment.

Participants' data will be taken from their medical records (charts), which were already collected as a part of their routine care between January 1, 2012, and January 1, 2022.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective, observational study of participants with Hereditary Angioedema with normal C1 esterase inhibitor (HAE) and Non-histaminergic Angioedema (NHAE) with normal C1-inhibitor function (nC1-INH) receiving various treatments between January 1, 2012, and January 1, 2022. The study will assess case numbers, treatments, outcomes, and healthcare resource utilization in the real-world setting.

This study will enroll approximately 90 to 150 participants. Participants will be enrolled in the following two cohorts:

* Participants with HAE nC1-INH
* Participants with NHAE nC1-INH

This study will have a retrospective data collection from January 1, 2012 to January 1, 2022 by using data from the participant medical charts that were already collected as part of routine care.

This multi-center trial will be conducted in Canada. The overall time for data collection in this study will be approximately 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥12 years of age with HAE nC1-INH or NHAE nC1-INH diagnosed by an HAE treating specialist based on some or all of the following:

1. Recurrent angioedema as documented by a healthcare professional within specialist charts
2. Normal C4
3. Normal C1 level and function
4. Condition worsened with estrogen if estrogen is/was being received
5. Lack of response to corticosteroid and high-dose regular and/or prophylactic antihistamine(s) treatment(s)
6. Family history of non-histaminergic angioedema for patients with HAE nC1-INH

Exclusion Criteria:

1. Other types of angioedema (type-1 HAE, type-2 HAE, acquired angioedema, etc.)
2. Not meeting the above diagnostic criteria for inclusion
3. Response to treatments used for histamine-related angioedema

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with confirmed diagnosis of HAE nC1-INH or NHAE nC1-INH prior to January 1, 2022.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants Diagnosed With HAE nC1-INH at Each Site | Up to approximately 10 years
Number of Participants Diagnosed With NHAE nC1-INH at Each Site | Up to approximately 10 years
Number of Participants Categorized by Type of Treatments Received by Participants | Up to approximately 10 years
Average Dose for Each Type of Treatment Received by Participants | Up to approximately 10 years
Average Duration of Treatment for Each Type of Treatment Received by Participants | Up to approximately 10 years
Number of Participants Categorized by Type of Settings Where Treatment was Received | Up to approximately 10 years
  Categories of treatment settings include: home, hospital, physician office, emergency room visits (ER), and other.
Number of Participants Receiving Multiple Long-Term Prophylaxis (LTP) Therapies at Once | Up to approximately 10 years
  Number of participants will be reported by number of LTP therapies received at once.
Number of Participants Receiving Multiple LTP Therapies Categorized by Combination and Order of Treatments Received | Up to approximately 10 years
Number of Attacks Occurring per Three-Months | Before and after initiation of treatment up to end of the study (up to approximately 10 years)
Number of Participants Categorized by Severity of Attack per Three Months | Before and after initiation of treatment up to end of the study (up to approximately 10 years)
  Categories of severity are planned to include ER, use of rescue medication(s), (%) intubation, hospitalization, and laryngeal involvement.
Number of Participants by Body Sites Affected by Attacks per Three Months | Before and after initiation of treatment up to end of the study (up to approximately 10 years)
  Body sites will include face, lip, tongue, gastrointestinal (GI) system, larynx, extremities, and other.
Number of Participants with Symptoms of the Attack | Up to approximately 10 years
Time from Treatment (On-demand Therapy) to Symptom Improvement/Resolution | Up to approximately 10 years
Number of Primary Care Visits per Year Associated With Management of HAE nC1-INH or NHAE nC1-INH | Up to approximately 10 years
Number of Walk-in Visits per Year Associated With Management of HAE nC1-INH or NHAE nC1-INH | Up to approximately 10 years
Number of Unscheduled Physician Visits per Year Associated With Management of HAE nC1-INH or NHAE nC1-INH | Up to approximately 10 years
Number of Emergency Room Visits per Year Associated With Management of HAE nC1-INH or NHAE nC1-INH | Up to approximately 10 years
Number of Hospitalizations per Year Associated With Management of HAE nC1-INH or NHAE nC1-INH | Up to approximately 10 years
Number of Intubations per Year Associated With Management of HAE nC1-INH or NHAE nC1-INH | Up to approximately 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- Canada (6):
  - Alberta Health Services, Calgary, Alberta
  - Alberta Health Services, Edmonton, Alberta
  - Vancouver Allergy Clinic, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Hamilton Health Science Corporation, Hamilton, Ontario
  - CHU de Québec - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/75ffe7820bc84741?idFilter=%5B%22TAK-743-4013%22%5D